CLINICAL TRIAL: NCT03729583
Title: The Effects of Breathing Retraining on Dyspnoea Measures and the Six-Minute Walking Distance in Patients With Interstitial Lung Diseases
Brief Title: The Effects of Breathing Retraining in Patients With Interstitial Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Melanie Axiak, Principal Investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAxiak
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group consisted of 15 patients with a diagnosis of ILD. They received a 12-week Pulmonary Rehabilitation (PR) programme without breathing retraining All patients were medically stable and referred by their caring respiratory consultant
  Interventions: Behavioral: Pulmonary Rehabilitation
- Active group (Experimental): The active group consisted of 15 patients with a diagnosis of ILD. They received a 12-week Pulmonary Rehabilitation (PR) programme with breathing retraining exercises. All patients were medically stable and referred by their caring respiratory consultant
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — A 12 week high intensity PR programme was delivered to both groups. The active group had additional breathing control interventions and exercises
  Other Names: Respiratory Rehabilitation

SUMMARY:
Breathing retraining has been reported to lead to improvements in dyspnoea and walking distance in chronic obstructive pulmonary disease (COPD) patients. Evidence regarding the effects of such an intervention in ILD patients is though lacking. In view of this, the aims of such a study were to identify whether breathing retraining led to better management of dyspnoea and improved walking distance in ILD patients.

DETAILED DESCRIPTION:
One of the commonest symptoms experienced in patients with a diagnosis of interstitial lung disease (ILD) is shortness of breath, a symptom which greatly affects their abilities to carry out activities of daily living. Breathing retraining has been reported to lead to improvements in dyspnoea and walking distance in chronic obstructive pulmonary disease (COPD) patients. Evidence regarding the effects of such an intervention in ILD patients is though lacking. In view of this, the aims of such a study were to identify whether breathing retraining led to better management of dyspnoea and improved walking distance in ILD patients. Twenty Seven ILD patients were randomly distributed to either the control group (n=15) which received a 12-week Pulmonary Rehabilitation (PR) programme without breathing retraining or the active group (n=12) which received a 12-week PR programme with breathing retraining. All patients had both the 6-minute walk test and their level of breathlessness assessed using the Dyspnoea Borg scale assessed at baseline and at 4 weekly intervals for a 12-week period throughout the programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of ILD and who were referred for PR

Exclusion Criteria:

* Patients who had musculoskeletal or neurological conditions affecting the outcome measures
* Patients who required oxygen therapy and did not accept administration
* Patients with unstable cardiovascular conditions
* Patients who were not willing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | Change in walking distance from baseline to 12weeks
  A walk test to examine exercise endurance

SECONDARY OUTCOMES:
Dyspnoea score | Change in dyspnoea measures from baseline to 12weeks
  Borg scale

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Axiak, BSc, Principal Investigator — University of Malta
Locations (1):
- Melanie Axiak, Mosta, Malta

IPD SHARING:
Plan to Share IPD: No
All data will be provided in the publication